CLINICAL TRIAL: NCT01488500
Title: Cardiovascular Effects of Experimental Exposure to Woodsmoke in Man
Brief Title: Woodsmoke Exposure and Cardiovascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Umeå University (Other)
Responsible Party: Principal Investigator, Jeremy Langrish, Clinical Lecturer and Specialty Registrar in Cardiology, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: WOODSMOKE II
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Respiratory Inflammation; Systemic Inflammation
Keywords: Wood smoke; inflammation; lung function; arterial stiffness; heart rate variability; Respiratory and systemic inflammation following exposure to woodsmoke in healthy volunteers
MeSH Terms: conditions — Inflammation | interventions — Bronchoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Filtered air exposure (Experimental): 3 hour exposure to filtered air with intermittent exercise
  Interventions: Other: Bronchoscopy
- Wood smoke exposure (Experimental): 3 hour exposure to dilute wood smoke generated from incomplete combustion in a wood burning stove at approximately 300 mcg/m3
  Interventions: Other: Bronchoscopy
- Wood pellet smoke emission (Experimental): 3 hour exposure to dilute wood smoke generated from wood pellets during incomplete combustion during intermittent exercise at approximately 300 mcg/m3
  Interventions: Other: Bronchoscopy

INTERVENTIONS:
Other: Bronchoscopy — 24 hours after exposure, a bronchoscopy will be performed to allow analysis of cells and inflammatory markers in bronchial wash, bronchioalveolar lavage and lung biopsies.

SUMMARY:
Air pollution is linked to respiratory and cardiovascular disease. Wood smoke is a common air in many parts of the world and previous studies indicate that wood smoke induce oxidative stress in the respiratory tract. It is not determined how different types of biomass combustion affect human health. In this study the investigators plan to investigate how inhalation of wood smoke and pellets smoke affect respiratory and cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Use of regular medication except the oral contraceptive pill
* Current smokers
* Significant occupation exposure to air pollution
* Intercurrent illness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Respiratory inflammation | 24 hours after exposure to air or woodsmoke
  Bronchoscopy will be performed, and samples collected by bronchoalveolar lavage and bronchial biopsy. Samples will be analysed for cell counts, histology and inflammatory markers.

SECONDARY OUTCOMES:
Central arterial stiffness | Baseline and for 1 hour after exposure
  Central arterial stiffness will be measured at baseline and for the 1 hour following the exposure using the SphygmoCor and Vicorder devices
Heart rate variability | 24 hours after the exposure
  Continuous electrocardiograms will be recorded using a holter monitor to determine heart rate variability
Systemic inflammation | 24 hours after the exposure
  Blood samples will be taken at intervals following the exposure to woodsmoke to measure circulating inflammatory markers
Lung function | Baseline and 24hrs after exposure
  Lung function will be assessed using spirometry before and after each exposure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Sandström, MD PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Sweden

REFERENCES:
- [Derived] Muala A, Rankin G, Sehlstedt M, Unosson J, Bosson JA, Behndig A, Pourazar J, Nystrom R, Pettersson E, Bergvall C, Westerholm R, Jalava PI, Happo MS, Uski O, Hirvonen MR, Kelly FJ, Mudway IS, Blomberg A, Boman C, Sandstrom T. Acute exposure to wood smoke from incomplete combustion--indications of cytotoxicity. Part Fibre Toxicol. 2015 Oct 29;12:33. doi: 10.1186/s12989-015-0111-7. PMID 26511835
- [Derived] Langrish JP, Watts SJ, Hunter AJ, Shah AS, Bosson JA, Unosson J, Barath S, Lundback M, Cassee FR, Donaldson K, Sandstrom T, Blomberg A, Newby DE, Mills NL. Controlled exposures to air pollutants and risk of cardiac arrhythmia. Environ Health Perspect. 2014 Jul;122(7):747-53. doi: 10.1289/ehp.1307337. Epub 2014 Mar 25. PMID 24667535
- [Derived] Unosson J, Blomberg A, Sandstrom T, Muala A, Boman C, Nystrom R, Westerholm R, Mills NL, Newby DE, Langrish JP, Bosson JA. Exposure to wood smoke increases arterial stiffness and decreases heart rate variability in humans. Part Fibre Toxicol. 2013 Jun 6;10:20. doi: 10.1186/1743-8977-10-20. PMID 23742058